CLINICAL TRIAL: NCT02401789
Title: Dimensional Alterations of the Edentulous Ridge Following Removal of Multiple Adjacent Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute Franci (Other)
Responsible Party: Principal Investigator, Cecchinato Denis, Dimensional alterations of the edentulous ridge following removal of multiple adjacent teeth., Institute Franci
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIS-D 2013-017
Record Dates: First submitted 2015-03-16; First posted 2015-03-30 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Multiple Adjacent Teeth; Bone Remodelling
Keywords: oral surgery; Implantology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- test - implant placement (Experimental): The possibility of counteracting unfavourable ridge modelling after multiple tooth extractions by placing implants in the fresh extraction sites
  Interventions: Device: Implants (OsseospeedTM,EV Astra Tech System, DentsplyTM, Mölndal)
- control- natural healing (No Intervention)

INTERVENTIONS:
Device: Implants (OsseospeedTM,EV Astra Tech System, DentsplyTM, Mölndal)
  Arms: test - implant placement

SUMMARY:
The objective of the present study is to evaluate if loss of multiple adjacent teeth will cause proportionally greater tissue diminution than the loss of single teeth the possibility of counteracting unfavourable ridge modeling after multiple tooth extractions by placing implants in the fresh extraction sites soft tissue alterations at implants and adjacent teeth

DETAILED DESCRIPTION:
The study will be designed as a prospective, randomized, controlled multicenter study evaluating the potential of endosseous implants (OsseospeedTM,EV, Astra Tech System, DentsplyTM, Mölndal, Sweden) placed in fresh extraction sockets to preserve the ridge dimensions at the edentulous site.

Three centers will be involved in the study namely, (i) Department of Periodontology, University of Padova, Italy, (ii) Institute Franci, Padova, Italy, (iii) Department of Periodontology, Sahlgrenska Academy, University of Gothenburg, Sweden.

Prior to the start of the study the human review board at the treatment centers must approve the study protocol as well as the informed consent forms.

Group assignment

Following the removal of the target teeth, the subject (site) will be randomly assigned to one of 2 groups:

Test group 1:

Implants (OsseospeedTM,EV Astra Tech System, DentsplyTM, Mölndal) will be used. Preparation of the osteotomy for the implant sites will include the use of drills. A guide drill will establish the buccal-palatal/lingual and mesio-distal position of the implants. The final osteotomy preparation will be done by a single pass of an appropriate drill. Using a handpiece at 20 rpms and 50 Ncm of torque the implant will be placed. Primary stability must be obtained. Furthermore, the operator must ensure that a blood clot properly fills the void in the fresh extraction sockets. A MucograftTM membrane (Geistlich Pharma, Wolhusen, Switzerland) will be adapted to the entrance of the hard tissue defects. Sutures will be placed to secure the position of the membrane.The treatment should follow the guidelines described in the Astra Tech Manuals 'Surgical Procedures' and 'Cement-or screw- retained restorations -Clinical and laboratory procedures'. To avoid excessive loading of the implant during the healing period, the patient is not allowed to use any implant supported temporary restorations.

After 4 months of healing abutments will be installed (Healing AbutmentTM or Healing Abutment ZebraTM). The soft tissue will be adapted and sutured back for a tight seal around the abutment. The restorative procedure will commence and the prosthetic device inserted.

Control group:

No material will be placed in the socket. A MucograftTM membrane (Geistlich Pharma, Wolhusen, Switzerland) will be adapted to the entrance of the hard tissue defects. Sutures will be placed to secure the position of the membrane. After 4 months of healing implant installation will take place (see above) and after another 3 months the prosthetic rehabilitation will be performed.

Follow-up period During a 3 year follow-up period the subjects of the test and control groups will be recalled every 6 months for professional tooth cleaning.

Procedures:

Stone models:

An impression of the target sites using a polyphosphate-based impression material will be taken prior to tooth extraction and a stone model of the extraction site and adjacent teeth will be produced.

New impressions and stone models will be produced one week following tooth extraction and after 4 months of healing and after 1,2 and 3 years of follow-up.

Radiographs:

The supra-gingival portion of the teeth in (a duplicate of) the stone model (see above) to be extracted will be carefully removed. The center of the future "extraction sites" will be identified. A rigid acrylic splint - a guide including a quartz marker (Dual Scan MarkerTM ( Materialize Dental NV, Leuven, Belgium)- will be produced. This guide will be used for the CBCT scans.

Immediately after a careful flapless extraction of the teeth, (i) a cone beam computerized tomographic (CBCT) examination of the edentulous sites will be performed. The radiographic examination will be performed with the Planmeca ProMax3D unit (Planmeca Oy, Helsinky, Finland). The images will be acquired by means of the Planmeca Romexis software and processed by a computer. Acquisition will be performed for 24s (volumetric dimension of 8 x 8 cm) with the Planmeca tomography acquisition protocol: voxel size: 0.15 mm; Grey scale: 12 bits; focal spot: 0.5x0,5 mm; image detector: amorphous silicon flat panel; image acquisition: single 270° rotation. The images will be generated in DICOM format and the files of each patient will be saved and analyzed.

(ii) a series of standard intraoral radiographs, using the paralleling technique will be obtained from each experimental socket and inter-dental bone.

A new set of CBCT scans will be obtained after 4 months of healing following tooth extraction and after 3 year. New intraoral radiographs will be obtained prior to and after tooth extraction, after 4 months of healing (before and after implant placement) and after 1, 2 and 3 years.

Recordings:

On the stone models (mm and mm2)

1. Maximum bucco-lingual width (mm) at midline of each extraction socket (see Schropp et al. 2003)
2. The location of the crest -in relation to defined reference points at the adjacent teeth- (i) next to adjacent teeth (mm) , (ii) at the center of each extraction socket (mm and mm2 ) and (iii) at the position of the "inter-implant/tooth papillae"(mm) In the CBCT scans measurements will be made at (i) the center of each extraction socket, (ii) between the sockets ("inter-dental septum") (iii) at the septum next to adjacent teeth Intraoral radiographs The changes in the crestal bone levels will be assessed and by measuring the distance (MBL) from a defined reference point on the implant (adjacent tooth surface) to the most coronal bone-to implant contact on the mesial and distal aspect of the implant/tooth. In the radiographs the MBL distance will be recorded to the nearest 0.1 mm using a magnifying (X7) lens.

Clinical examination This examinations will be performed at the visit of placement of the permanent restoration and after 1,2, and 3 years and include the following; Soft tissue inflammation: The condition of the mucosa/gingiva around all implants and adjacent teeth will be assessed at 4 surfaces (mesial, distal, buccal, palatal) using a periodontal probe. Inflammation in the soft tissue will be considered present when a site bleeds on gentle probing (BoP).

Papilla fill: The degree of soft tissue fill in the inter-implant and tooth-implant sites will be determined according to the criteria of the Papilla Index System (scores 0 - 4) described by Jemt (1997).

Soft tissue margin: The distance between the margin of the permanent restoration and the most apical level of the soft tissue margin will be measured at the buccal aspect of the implants as well as a corresponding distance at neighboring teeth. This so called "mucosal zenith" value will be measured with a periodontal probe and expressed in mm.

Statistical methods Clinical outcome variables: Main outcome variable will be the alteration following tooth extraction of horizontal and vertical dimensions of the edentulous ridge including both soft and hard tissues. Secondary outcome variables will be implant survival at 1, 2, 3 years, radiographic bone level and soft tissue change at implants/adjacent teeth and extraction defects.

Power calculation based on the detection of a difference of 3 mm in mean crest width difference between treatment groups, assuming a standard deviation of 3.0 mm (Schropp et al 2003), and with an alpha error defined to 0.05 and beta error to 0.20 (power 80%), revealed that 17 subjects in each treatment group will be required. Considering a 10% drop out, a total of 40 patients/teeth must be included.

For analysis of clinical efficacy, data from two slightly different analysis populations will be used, i.e. the Per Protocol (PP) and the All Patients Treated (APT) populations. The primary objective is to determine the alterations in the buccal and palatal aspects of the size of the defect dimensions at implant placement and after healing. Results will be presented by appropriate descriptive and inferential statistics. Continuous variables will be presented by means of number of observations (N), minimum (min), median, maximum (max), mean and standard deviation (std). Discrete variables will be presented by frequency and percentage.

Experimental Schedule

Test group 1

Visit 1:

Soft tissue: all approximal surfaces (inflammation; PPD and Papilla Index) Impression: 2 stone models, preparation of Rx guide (stent) Rx: intra-oral radiograph(s)

Visit 2:

Extraction of target teeth, implant placement (non-submerged), wound closure, Mucograft membrane. Impression: stone model Rx: CBCT Visit 3: 4 months Abutment connection Visit 4: 5 months Placement of definitive restoration Soft tissue: all approximal and buccal surfaces (inflammation; PPD and Papilla Index) Rx: intra-oral radiographs and CBCT Visit 5: 1 year Soft tissue: all approximal and buccal surfaces (inflammation; PPD and Papilla Index) Rx: intra-oral radiographs and CBCT Visit 6 : 2 years Soft tissue: all approximal and buccal surfaces (inflammation; PPD and Papilla Index) Rx: intra-oral radiographs Visit 7 : 3 years Soft tissue: all approximal and buccal surfaces (inflammation; PPD and Papilla Index) Rx: intra-oral radiographs and CBCT

control group

Visit 1:

Soft tissue: all approximal surfaces (inflammation; PPD and Papilla Index) Impression: stone models, preparation of Rx guide (stent) Rx: intra-oral radiographs

Visit 2:

Extraction of target teeth, wound closure, Mucograft membrane Impression: stone model Rx: intra-oral radiographs, and CBCT Visit 3: 4 months Impression: stone model Rx: intra-oral radiographs, and CBCT Implant placement Visit 4: 7 months Abutment connection, Placement of definitive restoration Visit 5: 8 months Soft tissue: all approximal and buccal surfaces (inflammation; PPD and Papilla Index ) Rx: intra-oral radiographs and CBTC Visit 6, 7, 8 : 1 year, 2 years, 3 years

Soft tissue:

all approximal and buccal surfaces (inflammation; PPD and Papilla Index) Rx: intra-oral radiographs At visit 8 In addition Rx: CBTC

ELIGIBILITY:
Inclusion Criteria:

* presence of an intact extraction socket following removal of the natural teeth defined by: a marginal dehiscence defect of the facial bone wall of < 3 mm no facial fenestration present apical of the marginal bone crest

Exclusion Criteria:

* Untreated rampant caries and uncontrolled periodontal disease Uncontrolled diabetes or any other systemic or local disease or condition that would compromise post-operative healing Unable or unwilling to return for follow-up or unlikely to be able to comply with study procedures according to investigators judgement.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01; Primary Completion 2023-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Measurements of the change of the bone in between 2 or more teeth reported in millimeters after 6 month of the extraction in relation to the amount of the buccal-lingual reduction | 6 month.
Measurements of the change of the bone in between 2 or more teeth reported in millimeters after 6 month of the extraction in relation to the amount of the buccal-lingual reduction | 1 year
Measurements of the change of the bone in between 2 or more teeth reported in millimeters after 6 month of the extraction in relation to the amount of the buccal-lingual reduction | 2 year
Measurements of the change of the bone in between 2 or more teeth reported in millimeters after 6 month of the extraction in relation to the amount of the buccal-lingual reduction | 3 year
Measurements of the change of the bone in between 2 or more teeth reported in millimeters after 6 month of the extraction in relation to the amount of the buccal-lingual reduction | 4 year
Measurements of the change of the bone in between 2 or more teeth reported in millimeters after 6 month of the extraction in relation to the amount of the buccal-lingual reduction | 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- Franci Institute, Padua, Italy

REFERENCES:
- [Background] References Araújo, M, F Sukekava, J Wennström and J Lindhe (2006).